CLINICAL TRIAL: NCT02660853
Title: Exacerbations in Severe Asthma Patients: Mechanisms and Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13/LO/1198
Record Dates: First submitted 2015-11-02; First posted 2016-01-21 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Asthma
Keywords: Exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe Asthma (Other): Patients under Steps 4/5 of Asthma Treatment - SIGN (Scottish Intercollegiate Guidelines Network) / BTS (British Thoracic Society) Guidelines
  Interventions: Diagnostic Test: FEV1

INTERVENTIONS:
Diagnostic Test: FEV1 — Participants have FEV1 test

SUMMARY:
The purpose of this study is to investigate exacerbations in severe asthma with regard to symptoms, lung function, aetiology and biomarkers.

DETAILED DESCRIPTION:
Patients will be recruited from the Severe Asthma Clinics at Royal Brompton Hospital. At the first visit the investigators will enrol and characterise patients. This will involve asking patients to keep a diary record of PEFR(Peak Expiratory Flow Rate), spirometry, symptom scores, use of beta-agonist reliever and other treatments for 2 weeks. Bloods tests will be taken for markers of systemic inflammation. Markers of oxidative stress will be measured in blood, exhaled breath condensate (EBC) and urine: malondialdehyde (MDA) and 8-isoprostanes. Nitric oxide (NO) levels in exhaled breath will be measured measured twice daily for 2 weeks using a portable hand-held NO meter. If spontaneous sputum is not available, sputum will be induced using ultrasonic nebulization of isotonic saline. Profile of inflammatory cells, cytokines in supernatants, bacteriological culture and microbiome analysis will be measured in the sputum. Patients will be observed over 12 months during which time the number of exacerbations will be recorded on basis of objective measures with evaluation of ACQ (Asthma Control Questionnaire), daily morning and evening PEF (Peak Expiratory Flow). At the earliest onset of exacerbation, the patient will be requested to contact the Asthma Research Unit. Patients will then be asked to attend the laboratory where similar tests to the first visit will be performed. For other exacerbations not studied, the patient will be asked to keep a detailed diary record of symptoms with severity scoring and spirometric and PEF measurements (Exacerbation Diary) over a period of 2 weeks after onset of exacerbation.

As patients with severe asthma are usually very well experienced in what the symptoms of exacerbations are, they will therefore be asked to recognise their own exacerbations. Each patient has their own way of recognising an exacerbation and the investigators will discuss this with each patient and try and establish whether an earlier warning signal is possible. Patients will be asked to record their symptoms and lung function as soon as they feel the onset of an exacerbation, since exacerbations are recognised by the patient as events that are 'clinically identified by being outside the patient's usual range of day-to-day variation'. The patient will receive or administer treatments for the exacerbation as usual without interference from the Research Team except for starting any antibiotic therapies, which will be started (if prescribed) as soon as the visit studies have been completed. Those who have been hospitalized will not be studied, and only those who can attend the Clinical Research Unit will be studied.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be able to give informed consent. The definition of severe asthma will be on the basis of

  * Uncontrolled asthma: three or more of the following features present in any week in the previous 4 weeks:

    * Daytime symptoms more than twice per week
    * Any limitation of activities
    * Nocturnal symptoms once or more per week
    * Need for reliever treatment more than twice per week
    * Pre bronchodilator FEV1 <80% predicted or personal best OR
  * Frequent severe exacerbations (≥2 per year) OR
  * Require prescription of daily or alternate day oral corticosteroids (OCS) to achieve asthma control despite the prescription of high dose inhaled corticosteroids (>1000mcg fluticasone propionate daily or equivalent) or maintenance oral corticosteroids plus a long acting beta agonist or one other controller medication (for example anti-cholinergics, leukotriene receptor antagonists or theophylline).

Exclusion Criteria:

* • Current smoker, or Ex-smoker with a >10 year pack history or having smoked within the past 6 months

  * Significant alternative diagnoses that may mimic or complicate asthma, in particular dysfunctional breathing, panic attacks, and overt psychosocial problems (if these are thought to be the major problem rather than in addition to severe asthma)
  * Significant other primary pulmonary disorders in particular pulmonary embolism, pulmonary hypertension, interstitial lung disease and lung cancer
  * Subjects with emphysema and bronchiectasis should only be excluded if this is thought to be the major pulmonary disorder rather than in addition to severe asthma
  * Diagnosis or current investigation of occupational asthma
  * Any subjects currently participating, or having participated within 3 months of the first dose in a study using a new molecular entity, or the first dose in any other study investigating drugs.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian F Chung, MBBS MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Biomedical research Unit, Royal Brompton Hospital, Sydney Street, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Severe Asthma: Patients under Steps 4/5 of Asthma Treatment - SIGN (Scottish Intercollegiate Guidelines Network) / BTS (British Thoracic Society) Guidelines, Observational study
Period: Overall Study
Arm/Group | Severe Asthma
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Severe Asthma
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent Predicted FEV1
Description: From date of screening visit until date of first asthma exacerbation visit Percent predicted Forced Expiratory Volume in First Second
Time Frame: Baseline Visit, 12 months
Measure: Mean (Standard Deviation); unit: % of predicted value
Arm/Group | Severe Asthma
Number analyzed (Participants) | 25
% of predicted value
  baseline | 58.6 (20.4)
  During exacerbation | 56.3 (22.2)
Statistical Analysis 1: Comparison: Severe Asthma; Baseline versus during exacerbation; Test type: Superiority; p = 0.745, t-test, 2 sided

2. Secondary Outcome: Exhaled Breath Condensate
Description: pH and free Iron
Time Frame: Baseline Visit, 12 months
Population: No data collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

3. Secondary Outcome: Markers of Oxidative Stress in Urine
Description: malondialdehyde (MDA)
Time Frame: Baseline Visit, 12 months
Reporting Status: Not Posted, anticipated posting 2020-02

4. Secondary Outcome: Markers of Oxidative Stress in Urine
Description: 8-isoprostanes
Time Frame: Baseline Visit, 12 months
Reporting Status: Not Posted, anticipated posting 2020-02

5. Secondary Outcome: Sputum Analysis
Description: Eosinophils as percentage of total count
Time Frame: From baseline visit and 12 months
Population: Severe asthma at baseline
Measure: Mean (Standard Deviation); unit: Percentage of total sputum counts
Arm/Group | Severe Asthma
Number analyzed (Participants) | 25
Percentage of total sputum counts
  Baseline | 10.9 (30.6)
  At exacerbation | 4.47 (9.47)
Statistical Analysis 1: Comparison: Severe Asthma; Test type: Superiority; p = 0.326, t-test, 2 sided

6. Secondary Outcome: PCR for Respiratory Viruses
Description: nasopharyngeal swabs
Time Frame: Baseline Visit, 12 months
Population: No data collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

7. Secondary Outcome: Sputum Microbiome
Time Frame: Baseline Visit, 12 months
Population: No data collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

8. Secondary Outcome: Corticosteroid Insensitivity in Peripheral Blood Mononuclear Cells
Time Frame: Baseline Visit, 12 months
Population: No data collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

9. Secondary Outcome: Exhaled Nitric Oxide
Time Frame: Baseline Visit, 12 months
Population: Data were not collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

10. Secondary Outcome: Exhaled Hydrogen Sulphide
Time Frame: Baseline Visit, 12 months
Population: Data were not collected
Arm/Group | Severe Asthma
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Severe Asthma
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-06-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT02660853/Prot_SAP_ICF_000.pdf